CLINICAL TRIAL: NCT02819869
Title: The Combination Effect of Statin Plus Metformin on Relapse-free
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: insufficient for the fund
Sponsor: Taipei Medical University WanFang Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: N201510039
Record Dates: First submitted 2016-06-28; First posted 2016-06-30 (Estimated); Last update posted 2017-04-19 (Actual); Status verified 2016-10

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Hydroxymethylglutaryl-CoA Reductase Inhibitors

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Taking both statin and metformin Group (Experimental): The experimental group take Lotidon 500mg/ tablet per day and Lipitor 10mg/ tablet per day for two years or until of a recurrence.
  Interventions: Drug: Statin and Metformin use
- Non- taking both statin and metformin Group (No Intervention): Non- taking both statin and metformin.

INTERVENTIONS:
Drug: Statin and Metformin use
  Arms: Taking both statin and metformin Group

SUMMARY:
The study demonstrated that either statin or metformin served as notable use in reducing the incidence of many cancers.

DETAILED DESCRIPTION:
The study revealed the population-based cohort study investigated the protective effect of statin and metformin against cancer events in patients with HBV infection. The study demonstrated that either statin or metformin served as independent chemopreventive agents with a dose-response effect in reducing the incidence of cancer with a dose-response effect of the agents and an additive or synergistic effect of combining statin and metformin use in reducing the incidence of many cancers.1 And based on our data in animal models, administration of metformin and statin might enhance the therapeutic effect of local tumor through apoptotic and antiangiogenesis pathways. These results also seemed as the synergistic effect of statin and metformin combined use in tumor control.2 The aim of this study is to clarify the potential protective benefit of these drugs on the combination effect of Statin plus Metformin on relapse-free survival of HCC patients after local treatments in patients with HBV.

ELIGIBILITY:
Inclusion Criteria:

* 1. 20 years or older at the time of obtaining consent. 2. Systemic conditions are 0 to 2 score of Performance Status (according to Eastern Cooperative Oncology Group: ECOG). 3.Diagnosis of hepatocellular carcinoma is based on the following 1) or 2).

  1. Patients who are confirmed to have early tumor stain and typical finding(s) of hepatocellular carcinoma with CT or MRI imaging
  2. Patients who underwent tumor biopsy and are histopathologically diagnosed as hepatocellular carcinoma 4. First onset or recurrence of hepatocellular carcinoma is not more than 1 time.

  5. Patients who underwent the following 1) or 2) prior to registration to determine therapeutic effect.
  1. Patients who underwent local therapy to achieve complete hepatonecrosis and are confirmed to have complete hepatonecrosis with CT imaging or MRI.
  2. Patients who underwent surgical treatment(s) and are confirmed not to have residual tumor with CT or MRI imaging. 6. Patients who are given full explanation of study participation (including cancer notification) and submit written consent forms with their understanding as well as voluntary will for this study.

     Exclusion Criteria:

  <!-- -->

  1. Hepatocellular carcinoma: 1) Patients who have extrahepatic metastasis 2) Patients who have portal invasion 3) Patients who experienced with systemic administration of anti-malignant tumor drugs to treat hepatocellular carcinoma
  2. Patients with encephalopathy in which pharmacotherapy is ineffective
  3. Patients with ascites or pleural effusion that cannot be managed with diuretics
  4. Systemic conditions:

  <!-- -->

  1. Patients unable to receive oral administration
  2. Patients with a history of gastrectomy or extensive resection of digestive tract
  3. Patients who are suspected to have biliary occlusion, choleretic disorder,cholecystectomy, or malabsorption of liposoluble agents
  4. Patients with multiple cancers (within a 5-year cancer-free period [from the same day of 5 years earlier to the day of obtaining consent forms) 5. Drug administration:

  <!-- -->

  1. Patients on warfarin therapy
  2. Patients who already use statin or metformin 6.Other exclusion criteria

  <!-- -->

  1. Women of pregnant, lactating, childbearing potential, or with the intention of becoming pregnant
  2. Patients who are presently participating in another clinical study (except for follow-up surveys for study outcomes)
  3. Patients who are judged to be ineligible for study entry by the investigator or subinvestigator
  4. GOT or GPT three times greater than normal
  5. Cr. 1.5 times greater than normal
  6. Child-pugh score C

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2016-09-01 (Actual); Study Completion 2016-12-14 (Actual)

PRIMARY OUTCOMES:
relapse-free survival of hepatocellular carcinoma patients | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Fa-Moon Suk, bachelor, Study Director — Taipei Medical University, Taiwan, R.O.C.
Locations (1):
- Taipei Medical University - WanFang Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No